CLINICAL TRIAL: NCT01230814
Title: A Double-Blind, Randomized Trial of Monthly Treatment With Topical Metronidazole and Miconazole Co-formulated Vaginal Suppositories Versus Placebo for Preventing Vaginal Infections in HIV-seronegative Women
Brief Title: Topical Metronidazole and Miconazole Co-formulated Vaginal Suppositories for Preventing Vaginal Infections in HIV-seronegative Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-0070; DMID STI CTG 09-0070 PVI
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Bacterial Vaginosis; Candidiasis; Trichomoniasis
Keywords: Bacterial vaginosis, metronidazole, miconazole, vulvovaginal candidiasis, trichomonas vaginalis, women, Kenya
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis; Trichomonas Infections; Candidiasis, Vulvovaginal | interventions — Miconazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental): Intravaginal metronidazole 750 mg plus miconazole 200 mg (co-formulated suppositories) nightly for 5 consecutive nights each month; 117 Subjects.
  Interventions: Drug: Neo-Penotran® Forte (active ingredient Metronidazole & Miconazole Nitrate)
- Arm 2 (Placebo Comparator): Placebo suppositories nightly for five consecutive nights each month; 117 Subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neo-Penotran® Forte (active ingredient Metronidazole & Miconazole Nitrate) — Neo-Penotran® Forte (active ingredient Metronidazole & Miconazole Nitrate), co-formulated vaginal suppositories containing metronidazole 750 mg with miconazole 200 mg and excipients (Witepsol S 55). Witepsol S 55 is a hard fat suppository base. Such bases consist mainly of triglyceride esters of the higher saturated fatty acids along with varying proportions of mono- and diglycerides. 117 subjects receive nightly for 5 consecutive night each month.
  Arms: Arm 1
Drug: Placebo — Placebo vaginal suppositories, identical in appearance to the active product; contains Witepsol S 55, Titanium Dioxide and D+C yellow #10 with no metronidazole or miconazole.117 subjects receive nightly for 5 consecutive nights each month.
  Arms: Arm 2

SUMMARY:
This research study is about vaginal infections such as bacterial vaginosis, yeast infections, and trichomoniasis. Usually, these infections can be treated with medication, but sometimes they come back after treatment. Researchers want to know if using vaginal suppositories can decrease the risk of vaginal infections. Participants will include 234 women who are sexually active (greater than or equal to 4 episodes of sex with men during the past month), HIV-negative, 18 to 45 years old, with bacterial infection [vaginosis and/or vulvovaginal candidiasis (VVC) and/or Trichomonas vaginalis] detected by laboratory testing at a screening visit. Women will receive vaginal suppositories containing drug or inactive ingredients (placebo). Participation in the study will be about 12 months. Study procedures include: urine and blood tests, physical exams, and questionnaires.

DETAILED DESCRIPTION:
Vaginal infections including bacterial vaginosis (BV), vulvovaginal candidiasis (VVC), and Trichomonas (T.) vaginalis are common and have been associated with increased risk of HIV and other sexually transmitted infections (STIs) in multiple prospective studies. Effective interventions for prevention of vaginal infections could substantially reduce the risk of HIV and other STIs in women. A recently completed trial has demonstrated that monthly periodic presumptive treatment (PPT) can reduce vaginal infections and promote Lactobacillus colonization. However, the oral regimen of metronidazole 2 grams plus fluconazole 150 mg was not sufficiently effective to warrant moving to Phase III HIV/STI prevention trials using this intervention. The identification of more efficacious regimens for reducing vaginal infections is a crucial step towards the development of inexpensive, female-controlled, non-coitally dependent HIV/STI risk reduction interventions for women. There is growing evidence that higher doses and longer courses may be more effective for treatment of vaginal infections than single-dose therapy. The overall goal of this protocol is to conduct a randomized, double-blind, placebo-controlled trial to test the efficacy of monthly PPT with topical metronidazole 750 mg plus miconazole 200 mg (co-formulated suppositories) versus matching placebo suppositories nightly for five nights each month for reducing the rates of BV and VVC among HIV-seronegative women. This regimen could produce sufficient reductions in vaginal infections to support its use in Phase III HIV and STI prevention trials. The study participants will include 234 women who are sexually active (greater than or equal to 4 episodes of heterosexual intercourse during the past month), HIV-seronegative, 18 to 45 years old, with BV and/or VVC and/or T. vaginalis detected by laboratory testing at a screening visit. There will be two study arms. The treatment arm (117 subjects) will receive PPT with intravaginal metronidazole 750 mg plus miconazole 200 mg (co-formulated suppositories) for five consecutive nights each month. The placebo arm (117 subjects) will receive PPT with identical placebo intravaginal suppositories for five consecutive nights each month. Individual participants will be in the study for one year.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained and informed consent form (ICF) signed.
* Female, aged 18-45 years.
* Sexually active with greater than or equal to 4 episodes of sex with a male partner during the past month.
* Human immunodeficiency virus (HIV)-seronegative on both HIV tests in parallel screening.
* Presence of bacterial vaginosis (BV) and/or vulvovaginal candidiasis (VVC) and/or T. vaginalis infection at screening:

  1. BV: Microscopic criteria (Nugent's score greater than or equal to 7)
  2. VVC: Fungal elements (pseudohyphae, blastoconidia, or both) on vaginal saline wet mount plus a positive culture showing yeast on Sabouraud's agar.
  3. T. vaginalis infection: Identification of motile trichomonads on vaginal saline wet preparation.
* Able and willing to comply with study visit schedule and procedures during the 12-month period of follow-up.
* Able and willing to abstain from sex or to use non-latex condoms (provided) for 24 hours following insertion of each vaginal suppository.
* Willing to abstain from alcohol during, and for 48 hours after, treatment.
* Plan to remain in study area for the next year.
* Agree to not participate in other research studies involving drugs, medical devices, or vaginal products for the duration of study.

Exclusion Criteria:

* Currently pregnant (positive urine Beta-Human Chorionic Gonadotropin (hCG) or planning to conceive during the next 12 months (by self-report).
* Currently breastfeeding.
* Within first 3 months post-partum.
* Current menstruation - women who are currently menstruating may be enrolled following the completion of menses.
* History of 4 or more episodes of treatment for any vaginal infection in the past 12 months. This would be a cumulative total, including any treatment for bacterial vaginosis (BV) and/or vulvovaginal candidiasis (VVC) and/or Trichomonas vaginalis (TV) and/or syndromic.
* History of medical condition that would contraindicate use of the study product

  1. Porphyria
  2. Epilepsy
  3. Serious liver disease or signs and symptoms consistent with serious liver disease including jaundice, ascites, esophageal varices, encephalopathy, and bleeding disorders.
  4. Renal failure
* History of adverse reaction to the study medications (intravaginal metronidazole or miconazole).
* Current use of medication that may interact with the study drug (due to vaginal absorption of study drug)

  1. Warfarin
  2. Phenytoin
  3. Phenobarbital
  4. Disulfiram
  5. Cimetidine
  6. Lithium
  7. Astemizole
  8. Terfenadine
* Current use of oral or intravaginal antifungal medication.
* Current use of oral or intravaginal metronidazole, tinidazole, or clindamycin.
* Current use of latex diaphragm.
* As determined by the investigator, a medical condition or situation exists such that study participation would not be advisable.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States
- Kenya (3):
  - Women's Health Project - Ganjoni Municipal Clinic, Mombasa, Coast
  - University of Nairobi - Center for STD/HIV Research & Training, Nairobi, Nairobi County
  - University of Nairobi - Kenya AIDS Vaccine Initiative, Nairobi, Nairobi County

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Metronidazole Plus Miconazole: Intravaginal metronidazole 750 mg plus miconazole 200 mg (co-formulated suppositories) nightly for 5 consecutive nights each month.
- Arm 2: Placebo: Placebo suppositories nightly for five consecutive nights each month.
Period: Overall Study
Arm/Group | Arm 1: Metronidazole Plus Miconazole | Arm 2: Placebo
Started | 118 | 116
Completed | 105 | 112
Not Completed | 13 | 4
Not completed — Lost to Follow-up | 11 | 3
Not completed — Discontinued (not due to adverse event) | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Metronidazole Plus Miconazole | Arm 2: Placebo | Total
Number analyzed (Participants) | 118 | 116 | 234
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [24 to 34] | 29 [23 to 35] | 29 [24 to 34]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 117 | 115 | 232
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 116 | 234
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 118 | 111 | 229
  White | 0 | 4 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 118 | 115 | 233
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
  Kenya | 89 | 87 | 176

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Monthly Periodic Presumptive Treatment (PPT) Using Metronidazole With Miconazole Intravaginal Suppositories Versus Matching Placebo Nightly for Five Nights Each Month for Preventing Vulvovaginal Candidiasis (VVC).
Description: Percentage of follow-up visits (Months 2, 4, 6, 8, 10, 12) positive for VVC based on the presence of fungal elements (pseudohyphae, blastoconidia, or both) on vaginal saline wet mount plus a positive culture showing yeast on Sabouraud's agar.
Time Frame: Months 2, 4, 6, 8, 10, and 12.
Population: Intention to treat population which consisted of all women who were randomized and had at least one follow-up visit. Two women in the metronidazole with miconazole arm did not return after enrollment.
Measure: Number (95% Confidence Interval); unit: percentage of follow-up visits
Units Other Than Participants: Follow-up visits
Arm/Group | Arm 1: Metronidazole Plus Miconazole | Arm 2: Placebo
Number analyzed (Participants) | 116 | 116
Number analyzed (Follow-up visits) | 645 | 665
percentage of follow-up visits | 10.4 [8.2 to 13.2] | 11.3 [9.0 to 14.1]
Statistical Analysis 1: Comparison: Arm 1: Metronidazole Plus Miconazole vs Arm 2: Placebo; Each participant within a study arm was considered a cluster, with observations at a maximum of 6 visits. The percentage of visits at which VVC was detected was compared between metronidazole plus miconazole arm versus placebo arm using a chi-squared statistic adjusted for clustering using the method of Donner and Klar (2000); Test type: Superiority or Other; p = 0.690, Clustered chi-squared statistic — The a priori threshold for statistical significance for VVC was p<0.020 (two-sided); Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.62 to 1.37] — For the relative risk estimate, the metronidazole plus miconazole arm represented the numerator and the placebo arm represented the denominator such that a relative risk <1 indicates a lower percentage of positive test visits in the treated arm

2. Primary Outcome: Efficacy of Monthly Periodic Presumptive Treatment (PPT) Using Metronidazole With Miconazole Intravaginal Suppositories Versus Matching Placebo Nightly for Five Nights Each Month for Preventing Bacterial Vaginosis (BV).
Description: Percentage of follow-up visits (Months 2, 4, 6, 8, 10, 12) positive for BV as determined by applying standard microscopic scoring criteria (Nugent's criteria) to vaginal Gram stained slides. BV is diagnosed when the score is greater than or equal to 7.
Time Frame: Months 2, 4, 6, 8, 10, and 12.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of follow-up visits
Units Other Than Participants: Follow-up Visits
Arm/Group | Arm 1: Metronidazole Plus Miconazole | Arm 2: Placebo
Number analyzed (Participants) | 116 | 116
Number analyzed (Follow-up Visits) | 645 | 665
percentage of follow-up visits | 21.2 [18.0 to 25.1] | 32.5 [28.4 to 37.1]
Statistical Analysis 1: Comparison: Arm 1: Metronidazole Plus Miconazole vs Arm 2: Placebo; Each participant within a study arm was considered a cluster, with observations at a maximum of 6 visits. The percentage of visits at which BV was detected was compared between metronidazole plus miconazole arm versus placebo arm using a chi-squared statistic adjusted for clustering using the method of Donner and Klar (2000); Test type: Superiority or Other; p = 0.005, clutstered chi-squared statistic — The a priori threshold for statistical significance for BV was p<0.030 (two-sided); Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.48 to 0.87] — For the relative risk estimate, the metronidazole plus miconazole arm represented the numerator and the placebo arm represented the denominator such that a relative risk <1 indicates a lower percentage of test visits in the treated arm

3. Secondary Outcome: Efficacy of Monthly Periodic Presumptive Treatment (PPT) Using Metronidazole With Miconazole Intravaginal Suppositories Versus Placebo for Preventing Any Vaginal Infection (a Combined Endpoint Including BV, VVC, and Trichomonas Vaginalis Infection).
Description: Percentage of follow-up visits (Months 2, 4, 6, 8, 10, 12) positive for any of three vaginal infections (BV, VVC, Trichomonas vaginalis infection).
Time Frame: Months 2, 4, 6, 8, 10, and 12.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of follow-up visits
Units Other Than Participants: Follow-up visits
Arm/Group | Arm 1: Metronidazole Plus Miconazole | Arm 2: Placebo
Number analyzed (Participants) | 116 | 116
Number analyzed (Follow-up visits) | 645 | 665
percentage of follow-up visits | 32.6 [28.4 to 37.3] | 46.5 [41.6 to 51.9]

4. Secondary Outcome: Efficacy of Monthly Periodic Presumptive Treatment (PPT) Using Metronidazole With Miconazole Intravaginal Suppositories Versus Matching Placebo Nightly for Five Nights Each Month for Preventing BV by Clinical Criteria (Amsel's Criteria).
Description: Percentage of follow-up visits (Months 2, 4, 6, 8, 10, 12) positive for BV by clinical criteria (Amsel's criteria).
Time Frame: Months 2, 4, 6, 8, 10, and 12.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of follow-up visits
Units Other Than Participants: Follow-up visits
Arm/Group | Arm 1: Metronidazole Plus Miconazole | Arm 2: Placebo
Number analyzed (Participants) | 116 | 116
Number analyzed (Follow-up visits) | 645 | 665
percentage of follow-up visits | 14.4 [11.8 to 17.7] | 18.2 [15.2 to 21.7]

ADVERSE EVENTS:
Time Frame: Months 2, 4, 6, 8, 10, and 12, and any interim visits.
Description: Adverse events were followed until resolution even beyond the study-reporting period. Resolution of an adverse event is defined as the return to pretreatment status or stabilization of the condition with the expectation that it will remain chronic.
Arm/Group | Arm 1: Metronidazole Plus Miconazole | Arm 2: Placebo
Serious Adverse Events (participants affected / at risk) | 3/116 | 1/116
Other Adverse Events (participants affected / at risk) | 109/116 | 111/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Metronidazole Plus Miconazole (N=116) | Arm 2: Placebo (N=116)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Soft tissue injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Metronidazole Plus Miconazole (N=116) | Arm 2: Placebo (N=116)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 17 (21)
Abdominal pain lower (Gastrointestinal disorders) | 14 (17) | 9 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (25) | 11 (13)
Body tinea (Infections and infestations) | 8 (8) | 8 (10)
Chest pain (Cardiac disorders) | 8 (9) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 12 (16)
Dyspepsia (Gastrointestinal disorders) | 10 (13) | 13 (17)
Gastroenteritis (Gastrointestinal disorders) | 9 (10) | 7 (7)
Headache (Nervous system disorders) | 24 (31) | 36 (53)
Hypoaesthesia (Nervous system disorders) | 12 (17) | 12 (19)
Malaria (Infections and infestations) | 7 (10) | 9 (11)
Menorrhagia (Reproductive system and breast disorders) | 9 (9) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (15)
Nasopharyngitis (Reproductive system and breast disorders) | 6 (11) | 7 (9)
Nausea (Gastrointestinal disorders) | 5 (6) | 7 (9)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (8)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 18 (24)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 10 (11)
Soft tissue injury (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (5)
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (9)
Toothache (Gastrointestinal disorders) | 8 (9) | 8 (10)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 40 (64) | 36 (54)
Urinary tract infection (Renal and urinary disorders) | 14 (24) | 12 (13)
Vaginal discharge (Reproductive system and breast disorders) | 27 (55) | 43 (67)
Vaginal odour (Reproductive system and breast disorders) | 10 (19) | 5 (11)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 8 (13) | 6 (9)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 38 (62) | 44 (78)
Vulvovaginitis (Reproductive system and breast disorders) | 19 (23) | 19 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No